CLINICAL TRIAL: NCT02870764
Title: A Randomized, Double-blind, Placebo-controlled Trial of Dan-shen Extract in Patients With Stable Angina Pectoris
Brief Title: The Effect of Dan-shen Extract On Lipoprotein Associated PHospholipase A2 Levels IN Patients With Stable Angina Pectoris
Acronym: DOLPHIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Fourth People's Hospital (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, ChunLing Wang, Attending Doctor, Taizhou Fourth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TaizhouFPH-001
Record Dates: First submitted 2016-08-13; First posted 2016-08-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Angina, Stable; Inflammation
Keywords: Danshenduofensuanyan; Lp-PLA2; coronary artery disease; Salvia miltiorrhiza
MeSH Terms: conditions — Angina, Stable; Inflammation; Coronary Artery Disease | interventions — dan-shen root extract; salvianolic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dan-shen extract (Active Comparator): Based on the standard medical care, 200mg of Danshenduofensuanyan, added into 250ml of 0.9% saline injection, given by continuous IV infusion at 2.5ml/min within 2 hours, once a day during the patients' hospitalization. Danshen drop spill (30 pill/day) taken orally for 60 days after discharge.
  Interventions: Drug: Dan-shen extract; Other: Standard medical care
- Placebo (Placebo Comparator): Based on the standard medical care, placebo was 200mg of glucose, added into 250ml of 0.9% saline injection, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Drug: Placebo; Other: Standard medical care

INTERVENTIONS:
Drug: Dan-shen extract — A kind of injection made from a kind of Chinese herb: salvia miltiorrhiza
  Other Names: salvianolic acid; Depside salt from Salvia Miltiorrhiza; Danshen Dropping Pill; dropping salvia pill
  Arms: Dan-shen extract
Drug: Placebo — 200mg glugose added into 250ml 0.9% saline injection by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion.
  Arms: Placebo
Other: Standard medical care — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of Chronic Stable Angina (2007).

SUMMARY:
This is a randomized, double-blind, placebo-controlled, adaptive clinical trial, which will assess the effect of DanshenDuofensuanyan[Danshen (a kind of Chinese herbal drug) extract] treatment on Lipoprotein associated phospholipase A2 level in patients with stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 years-75 years;
2. Written informed consent;
3. Patients with a clinical diagnosis of chronic stable angina, which fulfil one of the following conditions:

   1. Symptoms that support the diagnosis of chronic angina and/or a history of an abnormal exercise response limited by angina and/or electrocardiograph (ECG) changes
   2. a history of myocardial infarction and ST-T changes,
   3. stenosis of more than 50 % in at least one major epicardial coronary artery, as shown by coronary angiography or computed tomography angiography,
   4. Coronary heart disease confirmed by radionuclide angiocardiography;
4. Patients with moderate angina pectoris, which is defined as Grade II or III on the Canadian Cardiovascular Society Angina Grading Scale.

Exclusion Criteria:

1. Patients with severe complications that would complicate the condition, as assessed by the investigator, including liver or renal dysfunction, severe cardiopulmonary dysfunction, pulmonary hypertension, chronic obstructive pulmonary disease, a history of epilepsy or cerebral haemorrhage.
2. Patients who were angina-free during the run-in period without taking any drug.
3. Patients who experienced myocardial infarction or who were classified as Grade IV on the Canadian Cardiovascular Society Angina Grading Scale within the preceding 3 months.
4. Patients with chest pain that is caused by any other disease (e.g., acute myocardial infarction, severe neurosis, menopausal syndrome or hyperthyroidism).
5. Patients with a history of drug-induced bleeding or a history of bleeding caused by warfarin.
6. Patients with a history of haematopoietic disorder.
7. Patients who have had surgery within the previous 4 weeks or who have a haemorrhagic tendency.
8. Women who are pregnant or lactating or who have a positive pregnancy test, or women who have a menstrual period at baseline.
9. Patients who are participating in other trials or who have participated in other trials within the past 3 months.
10. Patients with a history of allergy or with a known or suspected allergy to the study drug.
11. Patients with a known or suspected history of alcohol or drug abuse within the past 2 years.
12. Patients with a mental disorder.
13. Family members or relatives of the study centre staff.
14. Inability to adhere to study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Serum level of Lp-PLA2 | up to Day 60 after discharge

SECONDARY OUTCOMES:
The proportion of patients in each treatment group who had clinically significant change as defined by the angina-frequency score on the Seattle Angina Questionnaire | Day 0 and Day 60 after discharge
carotid arterial intima-media wall thickness | Day0 and Day 60 after discharge
Canadian Cardiovascular Society (CCS) grading of angina pectoris | Day 0 and Day 60 after discharge
Change in the electrocardiogram (EKG) | Day 0 and Day 60 after discharge
Changes in the Serum Lipid, the high-sensitivity C-Reactive Protein(hs-CRP) and the Platelet Aggregation Rate | Day 0 and Day 60 after discharge
Incidence of new-onset major vascular events | up to 60 days after discharge
  Major adverse vascular events include ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular-related death.
Incidence of severe hemorrhages | up to 60 days after discharge
  The definition of "Severe hemorrhages" is in accordance with the GUSTO bleeding criteria, including fatal intracranial hemorrhage (ICH), symptomatic intracerebral hemorrhage (sICH) or which could result in substantial hemodynamic compromise requiring treatment.
Incidence of moderate hemorrhages | up to 60 days after discharge
  The definition of "moderate hemorrhages" is in accordance with the GUSTO bleeding criteria, which requires blood transfusion but not results in hemodynamic compromise.

CONTACTS AND LOCATIONS:
Overall Officials: A'Di Chen, Master, Study Chair — Taizhou Fourth People's Hospital
Locations (1):
- Taizhou Fourth People's Hospital, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
We could provide individual participant data without leaking the patients' personal information if needed.

REFERENCES:
- [Background] Li B, Wang Y, Lu J, Liu J, Yuan Y, Yu Y, Wang P, Zhao X, Wang Z. Evaluating the effects of Danhong injection in treatment of acute ischemic stroke: study protocol for a multicenter randomized controlled trial. Trials. 2015 Dec 9;16:561. doi: 10.1186/s13063-015-1076-4. PMID 26654631
- [Background] Wang PQ, Li DD, Dong W, Liu J, Yu YN, Shen CT, Chen QG, Chen BW, Chen YD, Wang Z. Danhong injection in the treatment of chronic stable angina: study protocol for a randomized controlled trial. Trials. 2015 Oct 21;16:474. doi: 10.1186/s13063-015-0998-1. PMID 26489511
- [Background] Yao Y, Feng Y, Lin W. Systematic review and meta-analysis of randomized controlled trials comparing compound danshen dripping pills and isosorbide dinitrate in treating angina pectoris. Int J Cardiol. 2015 Mar 1;182:46-7. doi: 10.1016/j.ijcard.2014.12.112. Epub 2014 Dec 29. No abstract available. PMID 25585358
- [Background] Cheng TO. Cardiovascular effects of Danshen. Int J Cardiol. 2007 Sep 14;121(1):9-22. doi: 10.1016/j.ijcard.2007.01.004. Epub 2007 Mar 23. PMID 17363091
- [Background] Cai A, Li G, Chen J, Li X, Li L, Zhou Y. Increased serum level of Lp-PLA2 is independently associated with the severity of coronary artery diseases: a cross-sectional study of Chinese population. BMC Cardiovasc Disord. 2015 Feb 26;15:14. doi: 10.1186/s12872-015-0001-9. PMID 25879827
- [Background] White HD, Simes J, Stewart RA, Blankenberg S, Barnes EH, Marschner IC, Thompson P, West M, Zeller T, Colquhoun DM, Nestel P, Keech AC, Sullivan DR, Hunt D, Tonkin A; LIPID Study Investigators. Changes in lipoprotein-Associated phospholipase A2 activity predict coronary events and partly account for the treatment effect of pravastatin: results from the Long-Term Intervention with Pravastatin in Ischemic Disease study. J Am Heart Assoc. 2013 Oct 23;2(5):e000360. doi: 10.1161/JAHA.113.000360. PMID 24152981
- [Derived] Chen AD, Wang CL, Qin Y, Tian L, Chen LB, Yuan XM, Ma LX, Wang YF, Sun JR, Wang HS, Dai N; DOLPHIN investigator group. The effect of Danshen extract on lipoprotein-associated phospholipase A2 levels in patients with stable angina pectoris: study protocol for a randomized controlled trial - the DOLPHIN study. Trials. 2017 Dec 20;18(1):606. doi: 10.1186/s13063-017-2336-2. PMID 29262859